CLINICAL TRIAL: NCT06496256
Title: Randomized Trial of Barrigel® to Increase Distance Between the Rectum and Prostate Bed to Decrease Rectal Dose in Patients Receiving Moderately Hypofractionated Radiation Therapy Who Have Had Recurrence of Prostate Cancer After Prostatectomy
Brief Title: Barrigel® PPRT (Post-Prostatectomy Radiation Therapy) Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Palette Life Sciences, Inc. (Industry)
Collaborators: Teleflex (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0423-0001
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ultrasound, High-Intensity Focused, Transrectal

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled, single-blinded multicenter study
Who Masked: Participant
Masking Description: All subjects who sign a consent and meet inclusion and exclusion criteria will be randomized to the treatment or the control arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Treatment Arms (Experimental): Subjects will be injected Barrigel between the rectum and prostate bed using transrectal ultrasound for guidance.
  Interventions: Device: Barrigel; Device: Transrectal Ultrasound
- Control Arm (Sham Comparator): Subjects randomized to the control group will not receive Barrigel but will have a Transrectal ultrasound probe inserted to simulate that aspect of the injection of Barrigel.
  Interventions: Device: Transrectal Ultrasound

INTERVENTIONS:
Device: Barrigel — Barrigel is an absorbable gel based on Non-Animal Stabilized Hyaluronic Acid (NASHA™) that is injected into the peri-rectal space
  Arms: Treatment Arms
Device: Transrectal Ultrasound — All subjects will have a transrectal ultrasound (TRUS) conducted. In the control subjects this will act as a sham procedure. For the investigational subjects, the TRUS will be used to visualize the placement of the needle

SUMMARY:
Barrigel is intended to temporarily position the anterior rectal wall away from the prostate or prostate bed during radiotherapy treatment for prostate cancer and, in creating this space, it is the intent of Barrigel to reduce the radiation dose delivered to the anterior rectum.

DETAILED DESCRIPTION:
Barrigel is composed of biodegradable material and maintains space for the entire course of prostate or prostate bed radiotherapy and is intended to be absorbed by the patient's body over time.

To evaluate the safety and effectiveness of Barrigel to reduce the radiation dose delivered to the anterior rectum by creating a space when injected between the rectum and the prostate bed in men receiving definitive external beam radiation therapy (intensity-modulated radiation therapy) for recurrence of prostate cancer after radical prostatectomy.

A prospective, randomized, controlled, single-masked multicenter study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
3. Prostatectomy surgeon notes specifying successful bilateral nerve Sparing procedure
4. Documentation of an intra or interfascial radical prostatectomy
5. Confirmed diagnosis of adenocarcinoma of the prostate treated primarily with radical prostatectomy with pN0 or pNX pathologic stage
6. No radiographic evidence of local, regional, or distant metastatic disease via PSMA PET or Axumin fluciclovine F18 scan
7. Prostate specific antigen (PSA) 0.1 ng/mL or higher
8. Intent to receive definitive radiation therapy to the prostate bed
9. Written informed consent for study participation prior to study enrollment

Exclusion Criteria:

1. Known allergy to hyaluronic acid
2. Pathologic T4 disease
3. Prior local prostate cancer therapy including cryotherapy or brachytherapy.
4. Prior post-prostatectomy or pelvic radiation therapy
5. Planned elective pelvic lymph node radiation therapy
6. Prior anorectal surgery (e.g. low anterior resection, abdominoperineal resection, absence of a rectum)
7. Inflammatory bowel disease requiring treatment with steroids (e.g. Crohn's disease, ulcerative colitis)
8. Active connective tissue disorder including lupus or scleroderma
9. Any urogenital abnormality that could limit the ability to access the Barrigel injection site
10. White blood cell count <4000/uL or >12,000/uL.
11. Hemoglobin <10 g/dL (transfusion or other intervention to achieve this is acceptable).
12. Active bleeding disorder or clinically significant coagulopathy defined as PTT >35 seconds or INR >1.4 or platelet count <100,000/mm3.
13. Serum AST/ALT >2.5 times the institutional upper limit of normal
14. Creatinine >2.0 mg/dL
15. Bilirubin >2.0 mg/dL
16. History of chronic renal failure.
17. History of uncontrolled diabetes (e.g. symptomatic hyperglycemia that is not controlled with medical management; fasting blood glucose >300 mg/dL).
18. History of acquired immunodeficiency syndrome (AIDS). Patients with controlled HIV infection (CD4+ T-cell counts ≥ 350 cells/µL) and no history of AIDS-defining opportunistic infections may be included.
19. Contraindication to having an MRI or PSMA/PET scan (e.g. non-MRI compatible device).
20. Presence of bilateral hip implants, although unilateral hip implant may be permissible if the implant is MRI compatible and does not produce artifact that interferes with any requirements of the study protocol
21. Subject unable or unwilling to comply with study requirements
22. Any condition that in the investigator's opinion would prevent administration or completion of study therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction in volume of rectum receiving radiation dose | 3 months
  Investigational subjects only: Achievement of a ≥ 25% change in reduction in the volume of rectum receiving 90% of the prescription dose in 70% of the subjects.

SECONDARY OUTCOMES:
Grade 2 Toxicities | 3 Months
  Test whether the use of the Barrigel spacer does not increase the incidence of acute grade 2+ GI toxicity within the first 3 months, which will be assessed using the proportion of subjects who have one or more incidences of acute grade 2+ GI toxicity within the first 3 months.
Expanded Prostate Cancer Index Composite (EPIC) bowel QOL | 3 months
  Evaluate the change in Expanded Prostate Cancer Index Composite (EPIC) Bowel Assessment composite score (from baseline within 3 months after completion of radiation therapy. The EPIC is graded on a 12 point scale, with a higher score indicating a higher outcome.
Expanded Prostate Cancer Index Composite (EPIC) Urinary QOL | 3 months
  Evaluate the change in Expanded Prostate Cancer Index Composite (EPIC) Urinary Assessment composite score from baseline within 3 months after completion of radiation therapy. The EPIC is graded on a 12 point scale, with a higher score indicating a higher outcome.

OTHER OUTCOMES:
Adverse Events | 3 months
  All adverse events

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Summit Health, Clifton, New Jersey
  - Urology Austin, Austin, Texas
  - Houston Metro Urology, Houston, Texas
- GenesisCare Ringwood, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
Data will be submitted to FDA as part of a 510(k). Study data will be shared with other researchers for analysis and reporting after FDA clearance, including protocol, SAP, CSR, and raw data.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Within three months of the FDA decision.
Access Criteria: Qualified researchers with the intent to publish their results.